CLINICAL TRIAL: NCT01899001
Title: Improving Psychological Health and Cardiovascular Disease Risk in Women With PCOS
Brief Title: Mood and Nutrition Interventions in Polycystic Ovary Syndrome
Acronym: MANI-PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 818103
Record Dates: First submitted 2013-07-10; First posted 2013-07-15 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Polycystic Ovary Syndrome (PCOS)
Keywords: Polycystic Ovary Syndrome; PCOS; Depression; Anxiety; Weight loss; Exercise; Nutrition; Therapy; Mood symptoms; Stress
MeSH Terms: conditions — Polycystic Ovary Syndrome; Depression; Anxiety Disorders; Weight Loss; Motor Activity | interventions — Cognitive Behavioral Therapy; Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT and Nutrition Counseling (Experimental): 8 weeks of Cognitive Behavioral Therapy (CBT) and 16 weeks of Nutrition Counseling
  Interventions: Behavioral: Cognitive Behavioral Therapy; Behavioral: Nutrition Counseling
- Nutrition Counseling (Other): 16 weeks of Nutrition Counseling alone
  Interventions: Behavioral: Nutrition Counseling

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Participants will receive weekly, 30 minute sessions with a CBT-trained clinical psychologist for the first 8 weeks. Briefly, the purpose of CBT is to treat mood and associated anxiety disorders by changing dysfunctional thoughts that lead to negative mood states and maladaptive behaviors. Through the use of Socratic questioning, the therapist challenges the patient to observe the relationship between thoughts and feelings and to question the underlying beliefs that perpetuate negative affect. Ultimately, patients learns to recognize maladaptive automatic thoughts and develop a more rational and balanced way of thinking about themselves and the world around them.
  Other Names: CBT
  Arms: CBT and Nutrition Counseling
Behavioral: Nutrition Counseling — All women will receive nutrition/exercise counseling by a trained counselor. They will consume a self-selected diet of 1500-1800kcal/d of conventional foods based on the Food Guide Pyramid. Participants will also have an exercise goal that starts at 50 minutes per week and increases to 175 minutes per week. Sessions will teach standard weight loss skills, including self-monitoring, problem-solving, enlisting social support, and overcoming negative thoughts. Subjects will be asked to keep daily food intake and exercise logs which will be reviewed at the nutrition counseling sessions. These sessions will occur in person once weekly lasting on average 30 minutes for 16 sessions.
  Other Names: Dietary Counseling; Exercise Counseling

SUMMARY:
The purpose of this study is to help determine the best treatment plan for women with PCOS who are overweight or obese and experiencing significant symptoms of depression and anxiety.

Specifically, the investigators are attempting to see if there is a difference between cognitive behavioral therapy in combination with nutritional counseling in improving mood symptoms, response to stress, and risk factors for heart disease compared to nutrition counseling alone. The investigators hypothesize that combined treatment with Cognitive Behavioral Therapy (CBT) and nutritional counseling will be more beneficial.

DETAILED DESCRIPTION:
This study will assess the impact of treatment of mood and associated anxiety disorders in conjunction with nutritional/exercise counseling in overweight/obese women with PCOS on cardiometabolic risk. The investigators hypothesize that women with PCOS will have greater benefit from dual intervention (psychological and nutritional/exercise counseling) for change in depressive symptoms and cardiometabolic risk reduction compared to nutritional/exercise counseling alone. In addition, the investigators hypothesize that psychological counseling may improve cardiometabolic risk by decreasing stress responses and stress associated markers of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Polycystic Ovary Syndrome (PCOS)
* Overweight or obese (BMI 27-50)
* Screen positive for symptoms of depression

Exclusion Criteria:

* Smoking 5 or more cigarettes per day
* Severe depression/anxiety warranting immediate treatment
* Actively participating in a weight loss program
* Taking medications to control cholesterol or diabetes
* On hormonal therapy (must be discontinued to be eligible)
* Pregnancy or planning to become pregnant during the study period
* Inability to commute to Philadelphia for weekly study sessions

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-07; Primary Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Assess change in mood symptoms after Cognitive Behavioral Therapy (CBT) and nutritional/exercise counseling compared to nutritional/exercise counseling alone. | Baseline, Week 8, Week 16
  Changes in mood symptoms will be assessed using the CES-D, STAI, HRQOL

SECONDARY OUTCOMES:
Assess change in cardio metabolic risk factors after Cognitive Behavioral Therapy (CBT) and nutritional/exercise counseling compared to nutritional/exercise counseling alone. | Baseline, Week 8, Week 16
  Changes in cardio metabolic risk factors will be assessed using clinical parameters (blood pressure, waist circumference, BMI) and serum parameters (lipid profile, fasting glucose, insulin, total testosterone, free testosterone, sex hormone binding globulin, Apo A1, Apo B, hsCRP, IL-6)
Assess change in perceived stress and stress response after Cognitive Behavioral Therapy (CBT) and nutritional/exercise counseling compared to nutritional/exercise counseling alone. | Baseline, Week 8
  Changes in perceived stress and stress response will be assessed using the PSS and cortisol response to the Trier Social Stress Test (TSST)

CONTACTS AND LOCATIONS:
Overall Officials: Anuja Dokras, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn PCOS Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Dokras A, Clifton S, Futterweit W, Wild R. Increased risk for abnormal depression scores in women with polycystic ovary syndrome: a systematic review and meta-analysis. Obstet Gynecol. 2011 Jan;117(1):145-152. doi: 10.1097/AOG.0b013e318202b0a4. PMID 21173657
- [Background] Dokras A, Clifton S, Futterweit W, Wild R. Increased prevalence of anxiety symptoms in women with polycystic ovary syndrome: systematic review and meta-analysis. Fertil Steril. 2012 Jan;97(1):225-30.e2. doi: 10.1016/j.fertnstert.2011.10.022. Epub 2011 Nov 27. PMID 22127370
- [Background] Hollinrake E, Abreu A, Maifeld M, Van Voorhis BJ, Dokras A. Increased risk of depressive disorders in women with polycystic ovary syndrome. Fertil Steril. 2007 Jun;87(6):1369-76. doi: 10.1016/j.fertnstert.2006.11.039. Epub 2007 Mar 29. PMID 17397839
- [Background] Wild RA, Carmina E, Diamanti-Kandarakis E, Dokras A, Escobar-Morreale HF, Futterweit W, Lobo R, Norman RJ, Talbott E, Dumesic DA. Assessment of cardiovascular risk and prevention of cardiovascular disease in women with the polycystic ovary syndrome: a consensus statement by the Androgen Excess and Polycystic Ovary Syndrome (AE-PCOS) Society. J Clin Endocrinol Metab. 2010 May;95(5):2038-49. doi: 10.1210/jc.2009-2724. Epub 2010 Apr 7. PMID 20375205
- [Background] Kelly CC, Lyall H, Petrie JR, Gould GW, Connell JM, Sattar N. Low grade chronic inflammation in women with polycystic ovarian syndrome. J Clin Endocrinol Metab. 2001 Jun;86(6):2453-5. doi: 10.1210/jcem.86.6.7580. PMID 11397838
- [Background] Boulman N, Levy Y, Leiba R, Shachar S, Linn R, Zinder O, Blumenfeld Z. Increased C-reactive protein levels in the polycystic ovary syndrome: a marker of cardiovascular disease. J Clin Endocrinol Metab. 2004 May;89(5):2160-5. doi: 10.1210/jc.2003-031096. PMID 15126536
- [Background] Toulis KA, Goulis DG, Farmakiotis D, Georgopoulos NA, Katsikis I, Tarlatzis BC, Papadimas I, Panidis D. Adiponectin levels in women with polycystic ovary syndrome: a systematic review and a meta-analysis. Hum Reprod Update. 2009 May-Jun;15(3):297-307. doi: 10.1093/humupd/dmp006. Epub 2009 Mar 4. PMID 19261627
- [Background] Shroff R, Kerchner A, Maifeld M, Van Beek EJ, Jagasia D, Dokras A. Young obese women with polycystic ovary syndrome have evidence of early coronary atherosclerosis. J Clin Endocrinol Metab. 2007 Dec;92(12):4609-14. doi: 10.1210/jc.2007-1343. Epub 2007 Sep 11. PMID 17848406
- [Background] Rozanski A, Blumenthal JA, Kaplan J. Impact of psychological factors on the pathogenesis of cardiovascular disease and implications for therapy. Circulation. 1999 Apr 27;99(16):2192-217. doi: 10.1161/01.cir.99.16.2192. PMID 10217662
- [Background] Yusuf S, Hawken S, Ounpuu S, Dans T, Avezum A, Lanas F, McQueen M, Budaj A, Pais P, Varigos J, Lisheng L; INTERHEART Study Investigators. Effect of potentially modifiable risk factors associated with myocardial infarction in 52 countries (the INTERHEART study): case-control study. Lancet. 2004 Sep 11-17;364(9438):937-52. doi: 10.1016/S0140-6736(04)17018-9. PMID 15364185
- [Background] Ferketich AK, Schwartzbaum JA, Frid DJ, Moeschberger ML. Depression as an antecedent to heart disease among women and men in the NHANES I study. National Health and Nutrition Examination Survey. Arch Intern Med. 2000 May 8;160(9):1261-8. doi: 10.1001/archinte.160.9.1261. PMID 10809028
- [Background] Rutledge T, Linke SE, Krantz DS, Johnson BD, Bittner V, Eastwood JA, Eteiba W, Pepine CJ, Vaccarino V, Francis J, Vido DA, Merz CN. Comorbid depression and anxiety symptoms as predictors of cardiovascular events: results from the NHLBI-sponsored Women's Ischemia Syndrome Evaluation (WISE) study. Psychosom Med. 2009 Nov;71(9):958-64. doi: 10.1097/PSY.0b013e3181bd6062. Epub 2009 Oct 15. PMID 19834049
- [Background] Roest AM, Martens EJ, de Jonge P, Denollet J. Anxiety and risk of incident coronary heart disease: a meta-analysis. J Am Coll Cardiol. 2010 Jun 29;56(1):38-46. doi: 10.1016/j.jacc.2010.03.034. PMID 20620715
- [Background] Fagundes CP, Glaser R, Hwang BS, Malarkey WB, Kiecolt-Glaser JK. Depressive symptoms enhance stress-induced inflammatory responses. Brain Behav Immun. 2013 Jul;31:172-6. doi: 10.1016/j.bbi.2012.05.006. Epub 2012 May 22. PMID 22634107
- [Background] Kerchner A, Lester W, Stuart SP, Dokras A. Risk of depression and other mental health disorders in women with polycystic ovary syndrome: a longitudinal study. Fertil Steril. 2009 Jan;91(1):207-12. doi: 10.1016/j.fertnstert.2007.11.022. Epub 2008 Feb 4. PMID 18249398
- [Background] Azziz R, Marin C, Hoq L, Badamgarav E, Song P. Health care-related economic burden of the polycystic ovary syndrome during the reproductive life span. J Clin Endocrinol Metab. 2005 Aug;90(8):4650-8. doi: 10.1210/jc.2005-0628. Epub 2005 Jun 8. PMID 15944216
- [Background] Moran LJ, Pasquali R, Teede HJ, Hoeger KM, Norman RJ. Treatment of obesity in polycystic ovary syndrome: a position statement of the Androgen Excess and Polycystic Ovary Syndrome Society. Fertil Steril. 2009 Dec;92(6):1966-82. doi: 10.1016/j.fertnstert.2008.09.018. Epub 2008 Dec 4. PMID 19062007
- [Background] Wing RR, Epstein LH, Marcus MD, Kupfer DJ. Mood changes in behavioral weight loss programs. J Psychosom Res. 1984;28(3):189-96. doi: 10.1016/0022-3999(84)90019-9. PMID 6545356
- [Background] Galletly C, Moran L, Noakes M, Clifton P, Tomlinson L, Norman R. Psychological benefits of a high-protein, low-carbohydrate diet in obese women with polycystic ovary syndrome--a pilot study. Appetite. 2007 Nov;49(3):590-3. doi: 10.1016/j.appet.2007.03.222. Epub 2007 Apr 4. PMID 17509728
- [Background] Linden M, Zubraegel D, Baer T, Franke U, Schlattmann P. Efficacy of cognitive behaviour therapy in generalized anxiety disorders. Results of a controlled clinical trial (Berlin CBT-GAD Study). Psychother Psychosom. 2005;74(1):36-42. doi: 10.1159/000082025. PMID 15627855
- [Background] Felitti VJ, Anda RF, Nordenberg D, Williamson DF, Spitz AM, Edwards V, Koss MP, Marks JS. Relationship of childhood abuse and household dysfunction to many of the leading causes of death in adults. The Adverse Childhood Experiences (ACE) Study. Am J Prev Med. 1998 May;14(4):245-58. doi: 10.1016/s0749-3797(98)00017-8. PMID 9635069
- [Background] Cronin L, Guyatt G, Griffith L, Wong E, Azziz R, Futterweit W, Cook D, Dunaif A. Development of a health-related quality-of-life questionnaire (PCOSQ) for women with polycystic ovary syndrome (PCOS). J Clin Endocrinol Metab. 1998 Jun;83(6):1976-87. doi: 10.1210/jcem.83.6.4990. PMID 9626128
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Kirschbaum C, Pirke KM, Hellhammer DH. The 'Trier Social Stress Test'--a tool for investigating psychobiological stress responses in a laboratory setting. Neuropsychobiology. 1993;28(1-2):76-81. doi: 10.1159/000119004. PMID 8255414
- [Derived] Cooney LG, Milman LW, Hantsoo L, Kornfield S, Sammel MD, Allison KC, Epperson CN, Dokras A. Cognitive-behavioral therapy improves weight loss and quality of life in women with polycystic ovary syndrome: a pilot randomized clinical trial. Fertil Steril. 2018 Jul 1;110(1):161-171.e1. doi: 10.1016/j.fertnstert.2018.03.028. Epub 2018 Jun 13. PMID 29908771